CLINICAL TRIAL: NCT01222780
Title: Phase I Trial to Evaluate the Safety, Activity and Pharmacokinetics of Marqibo(Registered Trademark) (Vincristine Sulfate Liposomes Injection) in Children and Adolescents With Refractory Cancer
Brief Title: To Evaluate the Safety, Activity and Pharmacokinetics of Marqibo in Children and Adolescents With Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 100220; IND 59,056 (Registry Identifier: Talon Therapeutics); NCT01344850 (obsolete NCT alias)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Sarcoma; Neuroblastoma; Wilms Tumor; Leukemia; Lymphoma; Brain Tumors
Keywords: Hematologic Malignancies; Vincristine Sulfate; Maximum Tolerated Dose; Pharmacokinetics; Solid Tumors; Cancer; Pediatrics; Sarcoma; Wilms Tumor; Leukemia; Lymphoma; Brain Tumor
MeSH Terms: conditions — Sarcoma; Neuroblastoma; Wilms Tumor; Leukemia; Lymphoma; Brain Neoplasms; Hematologic Neoplasms; Neoplasms | interventions — Vincristine

STUDY DESIGN:
Intervention Model Description: Phase 1 Trial to Evaluate the Safety, Activity and Pharmacokinetics of Marqibo® (Vincristine Sulphate Liposomes Injection) in Children and Adolescents with Refractory Cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Marqibo (Experimental): Marqibo® (Vincristine sulfate liposomal) will be administered intravenously over 60 minutes (±10 minutes) every 7 days (±3 days) (Days 1, 8, 15, 22) for four doses (1 cycle). Cycles may be repeated every 28 days for a maximum of 6 cycles; additional cycles may be offered with evidence of acceptable toxicity and clinical benefit.
  * The trial follows a rolling phase I design with 2 to 6 subjects per dose level and standard definitions of MTD and DLT. At the MTD, a total of 6 additional subjects with relapsed or refractory ALL will be evaluated.
  * Detailed pharmacokinetic studies will be performed during the first treatment cycle
  Interventions: Drug: Marqibo

INTERVENTIONS:
Drug: Marqibo — Marqibo® intravenously (IV) over 60 minutes (+ 10 minutes) every 7 days (+ 3 days) for 4 consecutive weeks (day 1, 8, 15, 22) for a 28-day treatment cycle
  Other Names: Vincristin Sulfate Liposomal Injection

SUMMARY:
Background:

* Marqibo(Registered Trademark) is a new anticancer drug. It combines Vincristine sulfate, which is a widely used anticancer drug, and packages it into a tiny fat bubble known as a liposome. The goal of this is to improve the drug's ability to destroy cancer cells and help reduce the potential side effects of treatment.
* Vincristine sulfate was originally developed from chemicals found in the periwinkle plant and acts against multiple types of malignant cancer. It is approved for multiple cancer types including solid tumors and blood cancers.
* Research has shown that Marqibo(Registered Trademark) is able to slow or stop the growth of cancer cells in some adults, both alone and in combination with other chemotherapy drugs, but more research is needed to determine its use in children.
* There has been one previous small study of Marqibo(Registered Trademark) in children. Although some anti-cancer activity was seen, side effects and optimal dosing were not fully determined.
* As is seen with standard Vincristine suflate, the most common side effect of Marqibo(Registered Trademark) involves the nervous system. It can cause numbness and tingling in the hands and feet. Symptoms commonly improve when the drug is discontinued or the dose is lowered.

Objectives:

- To determine the safety and efficacy of Marqibo as a treatment for children who have been diagnosed with certain types of malignant cancer that has not responded to standard treatment.

Eligibility:

* Children and adolescents between 2 and 21 years of age who have been diagnosed with certain types of malignant cancer that has not responded to standard treatment.
* These cancer types include solids tumors, primary brain tumors, leukemias, and lymphomas.

DETAILED DESCRIPTION:
BACKGROUND

* Vincristine sulfate is a widely used antineoplastic agent of the alkaloid class of drugs derived from the periwinkle plant (Vinca rosea Linn.). It has activity against a wide number of malignancies. It is a cell-cycle-specific agent that arrests cell growth in the M-phase (metaphase) by binding specifically with tubulin and disrupting cell division. Its dose limiting toxicity (DLT) is virtually always neurological.
* Investigations over the past two decades have demonstrated that liposomal drug carriers are capable of increasing the therapeutic index of anticancer drugs by altering the drug s pharmacological behavior.
* Marqibo(Registered Trademark) is vincristine encapsulated in sphingomyelin/cholesterol (SM/CHOL) liposomes, developed to increase the activity of vincristine. It has been shown to have activity in Phase 2 studies in adults. Previous investigation of Marqibo(Registered Trademark) in children is limited. A small phase 2 study was conducted with dosing of 2.0mg/m2 every 14 days. The agent appeared to be well tolerated and some activity was seen, although data were quite limited.

OBJECTIVES

* To define the maximum tolerated dose (MTD), toxicity profile, dose-limiting toxicities, and pharmacokinetics in children and adolescents with solid tumors or hematologic malignancies receiving weekly intravenous doses of Marqibo(Registered Trademark).
* To define the tolerability and potential activity of Marqibo(Registered Trademark) in children and adolescents with relapsed or refractory acute lymphoblastic leukemia (ALL) at the pediatric MTD.

ELIGIBILITY

- Children and adolescents (greater than or equal to 2 years and < 21 years of age) with histologically confirmed relapsed or refractory malignant disease that is measurable or evaluable.

DESIGN

* Marqibo(Registered Trademark) will be administered intravenously over 60 minutes (+ or -10 minutes) every 7 days (+ or - 3 days) (Days 1, 8, 15, 22) for four doses (1 cycle). Cycles may be repeated every 28 days for a maximum of 6 cycles; additional cycles may be offered with evidence of acceptable toxicity and clinical benefit.
* The trial follows a standard phase I design with 3 to 6 subjects per dose level and standard definitions of MTD and DLT. At the MTD, a total of 6 additional subjects with relapsed or refractory ALL will be evaluated.
* Detailed pharmacokinetic studies will be performed during the first treatment cycle.

ELIGIBILITY:
* INCLUSION CRITERIA

AGE: Subjects must be greater than or equal to 2 years and < 21 years of age.

DIAGNOSIS: Histologically confirmed solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms tumor, hepatic tumors, germ cell tumors, and primary brain tumors. In subjects with brain stem or optic gliomas the requirement for histological confirmation may be waived.

-Histologically confirmed diagnosis of hematologic malignancy, including but not limited to acute lymphoblastic leukemia (ALL), acute myelogenous leukemia (AML), Hodgkin's lymphoma, and non-Hodgkin's lymphoma (NHL). Isolated CNS or testicular disease is NOT allowed.

MEASURABLE/EVALUABLE DISEASE: Subjects must have measurable or evaluable malignant disease.

PRIOR THERAPY:

* The subject s cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available to that subject at the time of study entry.
* Subjects must have had their last doses of therapy prior to receiving the first dose of the investigational agent as follows (provided there is complete recovery from any acute toxic effects of such):

  1. Chemotherapy at least 14 days (6 weeks for nitrosoureas);
  2. Radiation at least 21 days;
  3. Any investigational cancer therapy or monoclonal antibody therapy (e.g., rituximab) at least 30 days.

Exceptions to these requirements:

* Intrathecal chemotherapy: There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such.
* Radiation therapy: There is no time restriction in regard to prior radiation provided the volume of bone marrow treated is less than 10% and that there is measurable disease outside the radiation port.
* Patients receiving corticosteroids or hydroxyurea are eligible provided all of the following conditions are met.
* Patients with CNS tumors who are managed with steroids are eligible if they are on a stable or decreasing dose of steroids and have no worsening neurologic deficits for greater than or equal to 7 days prior to registration.
* The subject is not on both corticosteroids and hydroxyurea
* Corticosteroids are not being used to manage GVHD.
* There has been no increase in the hydroxyurea dose for 2 weeks prior to starting Marqibo.
* Subjects must have recovered from the toxic effects (Grade 1 or baseline) of all prior therapy before entry onto this trial.
* Subjects should be off hematopoietic colony stimulating factors for at least 72 hours prior to study entry.
* Subjects with prior history of stem cell transplantation must be off immunosuppressive therapy for at least 4 weeks and have no active graft-versus-host disease (GVHD) with the exception of Grade 1 acute at the time of entry onto this trial.

PERFORMANCE STATUS: Subjects have a performance level greater than or equal to 50.

HEPATIC FUNCTION: Subjects must have adequate liver function, defined as bilirubin < 2.0 times the upper limit of normal, SGPT (ALT) and SGOT (AST) < 2.5 times the upper limit of normal.

RENAL FUNCTION: Subjects must have an age-adjusted normal serum creatinine OR a creatinine clearance greater than or equal to 60 mL/min/1.73 m(2):

* For age less than or equal to 5 - Maximum Serum Creatinine: 0.8
* For age less than 5 or less than or equal to 10 - Maximum Serum Creatinine: 1.0
* For age less than 10 or less than or equal to 15 - Maximum Serum Creatinine: 1.2
* For age greater than 15 - Maximum Serum Creatinine: 1.5

INFORMED CONSENT/ASSENT: All subjects or their legal guardians (for subjects < 18 years of age) must sign a document of informed consent (POB eligibility screening protocol) prior to performing studies to determine subject eligibility. After confirmation of subject eligibility all subjects or their legal guardians must sign the protocol-specific informed consent to document their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (other than the studies that were performed to determine subject eligibility). Where deemed appropriate by the clinician and the child s parents or guardian, the child will also be included in all discussions about the trial and verbal assent will be obtained. The parent or guardian will sign the designated line on the informed consent attesting to the fact that the child has given assent.

DURABLE POWER OF ATTORNEY (DPA): Subjects who have brain tumors and who are 18 years of age will be offered the opportunity to assign a DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

BIRTH CONTROL: Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study. Females of childbearing potential must have a negative pregnancy test within 7 days prior to starting study drug.

ADDITIONAL INCLUSION CRITERIA FOR EXPANDED COHORT OF ACUTE LYMPHOBLASTIC LEUKEMIA (ALL) SUBJECTS

DIAGNOSIS: Subjects must have a diagnosis of relapsed or refractory ALL or lymphoblastic lymphoma with > 5% marrow blasts (M2 or M3). Isolated CNS or testicular disease is not allowed. If < 5% marrow blasts must have histologically confirmed leukemia in extramedullary organ(s).

EXCLUSION CRITERIA

Clinically significant unrelated systemic illness, such as uncontrolled serious infection or organ dysfunction, which in the judgment of protocol investigators would compromise the subject s ability to tolerate the investigational agent or interfere with the study procedures or results. This includes any condition or circumstance that in the opinion of the investigator would significantly interfere with the subject s protocol compliance and put the subject at increased risk.

CNS leukemia or lymphoma as manifested by any of the following:

* CSF WBC > 5/microL and confirmation of CSF blasts.
* Cranial neuropathies deemed secondary to underlying malignancy
* CT or MRI scan evidence.

  * Note: History of CNS involvement is not an exclusion criterion.
* Neutrophil count < 1,000/microL or platelet count of < 50,000/microL (except for the expanded ALL cohort, where there is no blood count requirement).
* Pregnant or breast-feeding females are excluded because Marqibo(Registered Trademark) may be harmful to the developing fetus or nursing child.
* Currently receiving other investigational agents.
* History of previously receiving Marqibo(Registered Trademark).
* History of allergic reactions or serious adverse events attributed to compounds of similar chemical or biologic composition to vincristine or components of Marqibo(Registered Trademark) (vincristine sulfate injection, sphingomyelin/cholesterol liposomes, sodium phosphate injection).
* Are eligible for stem cell transplantation. This implies that a suitable donor is readily available, that the primary oncology team and Principal Investigator recommend this as a preferred treatment option at the time of protocol evaluation, and that the subject is willing to undergo stem cell transplantation.
* Presence of preexisting Grade 2 or greater sensory or motor neuropathy.
* History of persistent greater than or equal to Grade 2 active neurologic disorders unrelated to chemotherapy.
* Positive for human immunodeficiency virus (HIV) due to the increased risk of complications.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Define the toxicity spectrum of Marqibo in children with cancer | up to 48 weeks
  Toxicity was graded according to the version 4.0 of the NCI Common Toxicity Criteria (CTCAE v4.0).
Determine of Marqibo® administered as a 60 minute intravenous infusion weekly (every 28 days constitute 1 cycle), in children and adolescents with refractory solid tumors and hematologic malignancies. | up to 48 weeks
  The MTD was defined as the dose level immediately below the dose level at which ≥2 subjects in a cohort of 2 to 6 subjects experienced a DLT.
Determine dose limiting toxicities (DLT) of Marqibo® administered as a 60 minute intravenous infusion weekly (every 28 days constitute 1 cycle), in children and adolescents with refractory solid tumors and hematologic malignancies. | up to 48 weeks
  DLT was graded according to the version 4.0 of the NCI Common Toxicity Criteria (CTCAE v4.0). Adverse events (AEs) that were considered disease-related (not suspected of relationship to Marqibo) were not considered dose-limiting toxicities. Only those AEs deemed suspected of a relationship to Marqibo were used in the definition of DLT.

SECONDARY OUTCOMES:
Evaluate the plasma pharmacokinetics of Marqibo in children with cancer. | 28 days
  PK samples were collected at cycle 1 before start of first infusion, 5 minutes post-infusion and at 1, 3, 6, 10, 24, 48, 72, 96, 120 and 144 hours (pre-dose #2 trough level). Area under the concentration time curve (AUC) to last measured time point after dose one was calculated via linear trapezoidal method and extrapolated to infinity (AUC0-∞) by adding the last plasma concentration after dose one divided by the rate constant, derived from the slope of the natural log-transformed concentrations and times on the terminal elimination phase of the concentration-time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Wayne, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ross JA, Olshan AF. Pediatric cancer in the United States: the Children's Oncology Group Epidemiology Research Program. Cancer Epidemiol Biomarkers Prev. 2004 Oct;13(10):1552-4. No abstract available. PMID 15466968
- [Background] Linabery AM, Ross JA. Trends in childhood cancer incidence in the U.S. (1992-2004). Cancer. 2008 Jan 15;112(2):416-32. doi: 10.1002/cncr.23169. PMID 18074355
- [Background] Chonn A, Cullis PR. Recent advances in liposomal drug-delivery systems. Curr Opin Biotechnol. 1995 Dec;6(6):698-708. doi: 10.1016/0958-1669(95)80115-4. PMID 8527843
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-C-0220.html